CLINICAL TRIAL: NCT04035330
Title: Effect of Using Etidronate in Sodium Hypochlorite Versus Sodium Hypochlorite Irrigating Solution on the Intensity of Postoperative Pain and Bacterial Load Reduction in Patients With Necrotic Pulp: A Randomized Clinical Trial
Brief Title: Effect of Etidronate in Sodium Hypochlorite Versus Sodium Hypochlorite on the Intensity of Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Laila Zakaria Ismail, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETID_NAOCL
Record Dates: First submitted 2019-07-21; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Necrotic Pulp
Keywords: etidronate; postoperative pain; bacterial load reduction; sodium hypochlorite irrigation
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative | interventions — Etidronic Acid; Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- etidronate in sodium hypochlorite (Experimental): It comes in a capsule containing 0.9 g of etidronate powder, which should be mixed immediately with 10 mL of a NaOCl solution of choice directly before treatment, resulting in a combined irrigant containing both active chlorine and approximately 9% etidronate. Irrigation with a total volume of 25 ml for each case
  Interventions: Combination Product: etidronate in sodium hypochlorite
- sodium hypochlorite (Active Comparator): irrigation with 2.5% NaOCl with a total volume of 25 ml for each case
  Interventions: Combination Product: sodium hypochlorite

INTERVENTIONS:
Combination Product: etidronate in sodium hypochlorite — using etidronate in sodium hypochlorite solution with a volume of 5 ml between each instrument to reach a total volume of 25 ml
  Arms: etidronate in sodium hypochlorite
Combination Product: sodium hypochlorite — irrigation with 25 ml 2.5% sodium hypochlorite . 5ml between each instrument.
  Arms: sodium hypochlorite

SUMMARY:
To compare the effect of using Etidronate in sodium hypochlorite versus sodium hypochlorite irrigating solution on:

* Postoperative pain in patients with necrotic pulp.
* Bacterial load reduction & main bacterial species detected preinstrumentation and post-instrumentaion
* Periapical Matrix metalloproteinase 9 level (MMP-9) postinstrumentation and pre-obturation

DETAILED DESCRIPTION:
Patients will be clinically and radiographically examined and their eligibility will be assessed Eligible patients will be treated in 2 visits

1. Anesthetizing the tooth using inferior alveolar nerve block technique by local anesthesia of 1.8 ml of 2% Mepivacaine with 1:100,000 epinephrine.
2. Removal of caries and/or coronal restorations completely with sterile bur and rubber dam will be applied.
3. Cleaning the operative field, including the tooth, the clamp, and rubber dam sheet, with 30% hydrogen peroxide until no further bubbling of the peroxide occurred. All surfaces will then be disinfected by a sterile cotton swab with a 5.25% sodium hypochlorite solution.
4. Preparation of access cavity using another sterile round carbide bur size 3 and Endo-z bur.
5. After completing the access, the operative field and the pulp chamber will be cleaned and disinfected once again in the same way mentioned above. NaOCl will be then neutralized with 5% sodium thiosulfate.
6. The patients will be randomly divided into 2 groups. Intervention group (9% Etidronate in 2.5% sodium hypochlorite root canal irrigant /Dual rinse) and control group (2.5% sodium hypochlorite root canal irrigant).
7. Confirming the patency of the root canals using stainless steel hand K-files size #10 and #15. Working length will be determined using an electronic apex locator then confirmed radiographically to be 1 mm shorter than radiographic apex. The canals to be enlarged to size #20.
8. The pre-instrumentation root canal sample (S1) as follows: a sterile paper point will be placed in the wider /largest canal to soak up the fluid in the canal with saline to a level approximately 1 mm short of the tooth apex based on diagnostic radiographs and estimated working length. The paper point will be left in the canal for at least 1 minute. Paper points will then be transferred aseptically to tubes containing 20 ml of sterile thioglycollate broth.
9. Mechanical preparation will be done using M PRO rotary files in an endodontic motor.The first file (18/.09) will be used as an orifice opener for two thirds of the working length followed by (20/.04) for the full working length and finally (25/.06). In-and-out motions will be applied with stroke lengths not exceeding 3 mm in the cervical, middle, and apical thirds until attaining the established working length. The first file is used with a continuous rotary motion at a speed of 500 rpm and torque of 3 Ncm. The second and third files are both used with a speed of 500 rpm and torque of 1.5 Ncm. The canal will be irrigated and recapitulated after the use of each instrument.
10. The canals will be thoroughly irrigated with the allocated irrigant (5ml for 1 min) using plastic disposable syringe with needle gauge 30 reaching 1 mm short of the working length. All teeth will receive the same volume of irrigant (25 ml)
11. The canal will then be dried by using sterile paper points and then flushed with 5 ml of 5% sodium thiosulfate followed by 5 ml distilled water to inactivate the NaOCl. The postinstrumentation sample (S2) will be taken from the canal as described above. In addition, the periapical sample (S3) will be collected after cleaning and shaping by introducing a fine sterile size 20 paper point 2 mm beyond the canal terminus for 1 min. This procedure was performed twice. The paper points were placed in a sterile micro-centrifugation tube (Merck) containing 2 mL of sterile physiological saline solution, and immediately transferred to a -80 °C freezer until further processing.
12. The access cavities will be closed using sterile cotton pellet and temporary filling and patients will be recalled after 1 week.
13. The patients will record their pain level on Visual analogue scale & Numerical rating scale at 6,12, 24 and 48 hours.
14. In the recall appointment after 1 week. Rubber dam will be applied and tooth will be disinfected as before. The previously sampled canal will be re-entered, flushing with saline and a second periapical sample (S4) will be taken. After the sampling, final flush with 2.5% NaOCL and 17% Ethylene diamine tetraacetic acid (EDTA) in the control group, and with 2.5% NaOCL and 9% Etidronate in the intervention group. Master cones of (0.40) taper gutta-percha will be fitted to the working length and a radiograph will be taken to ensure proper length. Obturation using resin-based root canal sealer. The access cavity will be restored with composite resin and occlusal contact will be checked.
15. The patients will be asked to record their pain level on VAS & NRS at 6, 12, 24 and 48 hours .
16. The details of the endodontic procedure for each patient will be recorded in the patient's procedure chart
17. Finally, the patient will be appointed after 48 hours to collect the outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic disease.
* Mandibular permanent premolar teeth:

  * Diagnosed clinically with pulp necrosis.
  * Absence of spontaneous pain
  * Slight widening in the periodontal membrane space or with a periapical radiolucency
* Patients' acceptance to participate in the trial.
* Patients who can understand pain scale and can sign the informed consent

Exclusion Criteria:

* Medically compromised patients: Pain levels and healing following treatment would be compromised as these patients have shown higher incidence of pain and lower healing rate.
* Pregnant women: Avoid radiation exposure, anesthesia, and medication.
* If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively might alter their pain perception.
* Patients reporting bruxism or clenching: Avoid further pressure on an already inflamed tooth inducing subsequent irritation and inflammation.
* Teeth that shows association with acute periapical abscess and swelling:

Need special treatment steps which could involve additional visits with incision and drainage. Also, it could influence initiation and progression of postoperative pain.

* Greater than grade I mobility or pocket depth greater than 5 mm. Need special surgical and/or periodontal therapy.
* Hopeless tooth.
* Vital teeth.
* Immature teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | upto 48 hours after 1st visit
  intensity of pain by Numerical rating scale from 0-10

SECONDARY OUTCOMES:
bacterial load reduction | 1 hour after root canal preparation
  pre and post instrumentation samples to count intracanal bacteria (CFU/ml)

OTHER OUTCOMES:
matrix metalloproteinase | one week after root canal preparation
  Periapical MMP-9 level will be determined by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Laila Z Ismail, M.Sc., Principal Investigator — Cairo University; Shaimaa I Gawdat, Ph.D, Study Chair — Cairo University; Randa El boghdadi, Ph.D, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morago A, Ordinola-Zapata R, Ferrer-Luque CM, Baca P, Ruiz-Linares M, Arias-Moliz MT. Influence of Smear Layer on the Antimicrobial Activity of a Sodium Hypochlorite/Etidronic Acid Irrigating Solution in Infected Dentin. J Endod. 2016 Nov;42(11):1647-1650. doi: 10.1016/j.joen.2016.07.023. Epub 2016 Sep 8. PMID 27616541
- [Background] Arias-Moliz MT, Ordinola-Zapata R, Baca P, Ruiz-Linares M, Garcia Garcia E, Hungaro Duarte MA, Monteiro Bramante C, Ferrer-Luque CM. Antimicrobial activity of Chlorhexidine, Peracetic acid and Sodium hypochlorite/etidronate irrigant solutions against Enterococcus faecalis biofilms. Int Endod J. 2015 Dec;48(12):1188-93. doi: 10.1111/iej.12424. Epub 2015 Jan 8. PMID 25515403
- [Background] Lottanti S, Gautschi H, Sener B, Zehnder M. Effects of ethylenediaminetetraacetic, etidronic and peracetic acid irrigation on human root dentine and the smear layer. Int Endod J. 2009 Apr;42(4):335-43. doi: 10.1111/j.1365-2591.2008.01514.x. Epub 2009 Feb 7. PMID 19220516
- [Background] Ballal NV, Gandhi P, Shenoy PA, Shenoy Belle V, Bhat V, Rechenberg DK, Zehnder M. Safety assessment of an etidronate in a sodium hypochlorite solution: randomized double-blind trial. Int Endod J. 2019 Sep;52(9):1274-1282. doi: 10.1111/iej.13129. Epub 2019 May 13. PMID 30993696
- [Background] Paque F, Rechenberg DK, Zehnder M. Reduction of hard-tissue debris accumulation during rotary root canal instrumentation by etidronic acid in a sodium hypochlorite irrigant. J Endod. 2012 May;38(5):692-5. doi: 10.1016/j.joen.2011.12.019. Epub 2012 Jan 23. PMID 22515905